CLINICAL TRIAL: NCT06237790
Title: A Comparative Analysis of Speech Perception Between Cochlear Implant Patients and DFNB9 Patients Receiving Gene Therapy
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023185-1
Record Dates: First submitted 2023-12-26; First posted 2024-02-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss; Genetic Disease; Speech Perception
Keywords: Congenital Hearing Loss; DFNB9; Gene Therapy; Cochlear Implant; Speech Perception
MeSH Terms: conditions — Hearing Loss; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gene Therapy Group: The study will recruit gene therapy patients who are definitely diagnosed with autosomal recessive deafness 9 (DFNB9).
- Cochlear Implant Group: The study will recruit cochlear implant patients with congenital deafness.

SUMMARY:
This cohort study aims to explore the trends and differences in multidimensional perceptual levels of patients after cochlear implants or gene therapy, as well as to comprehensively assess the efficacy of gene therapy for congenital deafness, thus providing a reference for making a well-rounded postoperative rehabilitation protocol for gene therapy patients.

DETAILED DESCRIPTION:
Cochlear implant patients exhibit improved speech perception in quiet environments after surgery, but their music perception and speech perception under noise are still unsatisfactory. Gene therapy is a novel and promising treatment for congenital hearing loss to recover natural hearing sensations. To date, for patients with congenital deafness, there has been no study on their ability to perceive and understand sounds, such as speech perception in noise, music and directional perception, after hearing recovery owing to gene therapy. In addition, the difference between the two treatments in those perceptual levels postoperatively remains unknown.

Therefore, the investigators designed a single-center cohort study. Based on the intervention method, congenital deafness patients are divided into two groups: the cochlear implant group and the gene therapy group. In the present study, a full-scale evaluation of the two groups will be conducted. The battery encompasses auditory speech perception, cognition, psychological status, and auditory cortex development. A comparative analysis will be conducted to examine multidimensional differences between the two groups, shedding light on the divergent outcomes of gene therapy and cochlear implants for patients with congenital deafness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital hearing loss with hearing thresholds ≥65 dB receive either gene therapy (previously received gene therapy and standardized postoperative rehabilitation and follow-up or plan to receive gene therapy), or cochlear implant surgery. Healthy participants with bilateral hearing thresholds within the normal range (≤20 dB), generally matched to the gene therapy group and the cochlear implant group by age and sex.
* Age ≥ 6 months old, regardless of gender.
* Mandarin Chinese as the native language.
* Participants and their guardians must provide informed consent before the trial, voluntarily sign a written consent form, and commit to follow-up at specified time points.
* Capable of effective communication with researchers under the guardian's assistance and willing to cooperate and comply with the researchers' requirements.
* The participant's guardians should have a correct understanding of the trial and appropriate expectations regarding potential benefits.

Exclusion Criteria:

* Presence of other otological disorders that may interfere with the surgical outcome or interpretation of study endpoints, such as middle/inner ear dysplasia or malformations that affected the therapeutic effect revealed in CT/MRI scans within 3 months, vestibular-cochlear nerve abnormalities, acute/chronic otitis media, Meniere's disease, etc.
* Presence of other severe congenital diseases.
* Presence of severe systemic diseases or in the acute onset of diseases, such as pulmonary tuberculosis, active hepatitis B or C infection, active herpes zoster infection, pancreatitis, renal insufficiency, etc.
* Individuals with low immunity, a history of immune deficiency or organ transplantation.
* Individuals with a history of neurological or mental disorders, such as epilepsy or dementia.
* Patients with contraindications for surgery or anesthesia assessed by a surgeon, anesthetist, or designated personnel, such as cardiovascular or cerebrovascular events in the past 6 months, allergies to the planned medications, etc.
* Gene therapy group: gene therapy did not restore hearing; Cochlear implant group: presence of hereditary syndromic deafness or other conditions that seriously affect the efficacy evaluation.
* Any other conditions for which the investigators consider the subject unsuitable for participation in this clinical study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The number of enrollments in the gene therapy group is expected to be 90, and that of the cochlear implant group is expected to be at least 90, according to the pairing ratio of at least 1:1 between the cochlear implant group and gene therapy group. An estimated 30 healthy subjects are expected to be recruited (optional, subject to recruitment feasibility) for electroencephalography and/or functional near-infrared spectroscopy assessments.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Meaningful Auditory Integration Scale (MAIS)/Infant-toddler Meaningful Auditory Integration Scale (IT-MAIS): the MAIS (≥3 years old)/IT-MAIS (0~3 years old) is an auditory perception test with a total score of 40 points. The higher the score the better the hearing ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Categories of Auditory Performance (CAP): the CAP is an auditory perception test with a total levels of 8. The higher the level the better the hearing ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Speech Intelligibility Rating (SIR): the SIR is a speech perception test with a total levels of 5. The higher the level the better the hearing ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Meaningful Use of Speech Scale (MUSS): the MUSS is a speech perception test with a total score of 50 points. The higher the score the better the hearing ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Speech, Spatial, and Other Qualities of Hearing Scale for Parents (SSQ-P): the SSQ-P is an auditory speech and sound location perception test with a total score of 10 points. The higher the score the better the auditory speech and sound location ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  Mandarin Speech Perception (MSP): the MSP is a speech test software included the perception tests of monosyllable, disyllable and sentence recognition in quiet and noise environment. The higher the score the better the auditory speech ability.
Auditory speech perception | Preoperation, week 13, week 26 and week 52
  The Angel Test: the Angel Test is a speech test software included the perception tests of environmental sound test, final recognition test, initial recognition test and lexical tone test in quiet environment. The higher the score the better the auditory speech ability.

SECONDARY OUTCOMES:
Cognitive function | Preoperation, week 13, week 26 and week 52
  Griffiths development scales(GDS)/Wechsler Intelligence Scale for Children, 4e (WISC-IV): the GDS (0~6 years old)/WISC-IV (7~16 years old) is a cognitive function test. The higher the score the better the cognitive function.
Psychological status | Preoperation, week 26 and week 52
  Strengths and Difficulties Questionnaire(SDQ): the SDQ is a psychological status test with a total score of 25 points. The lower the score the better the psychological status.
Auditory cortex development | Preoperation, week 13, week 26 and week 52
  Electroencephalogram (EEG): the EEG is a non-invasive brain imaging method that uses brain maps to assess changes in auditory and speech-related cortex.
Auditory cortex development | Preoperation, week 13, week 26 and week 52
  Functional near-infrared spectroscopy (fNIRS): the fNIRS is a non-invasive brain imaging method that uses brain maps to assess changes in auditory and speech-related cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Yilai Shu, M.D. & Ph.D., Study Chair — Eye & ENT Hospital of Fudan University
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No